CLINICAL TRIAL: NCT03972644
Title: Danish National Randomized Study on Early Aortic Valve Replacement in Patients With Asymptomatic Severe Aortic Stenosis
Acronym: DANAVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Jordi Dahl, Associate Professor, MD, Ph.D., Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20190006
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Aortic Valve Stenosis; Diastolic Dysfunction
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early intervention (Active Comparator): Patients will undergo aortic valve replacement immediately
  Interventions: Procedure: Aortic valve replacement
- Watchfull waiting (No Intervention): Patients will be followed and treated as recommended by guidelines.

INTERVENTIONS:
Procedure: Aortic valve replacement — Open heart surgery or transcatheter surgery
  Arms: Early intervention

SUMMARY:
The purpose of this study is to examine the impact of early surgery in patients with asymptomatic severe aortic valve stenosis with signs of subclinical LV dysfunction despite preserved LVEF, with a watchfull waiting approach.

DETAILED DESCRIPTION:
Since the seminal paper by Ross and Braunwald, the development of symptoms has been regarded as one of the most important precursors of a poor outcome in aortic stenosis (AS), and is today half a century later, still the leading reason for referral for aortic valve replacement (AVR). The development of symptoms is however often preceded by structural changes in the left ventricle (LV).These changes including concentric remodeling and LV hypertrophy have been regarded as compensative measures to adapt the LV to increased ventricular afterload. Although LV hypertrophy may preserve wall-stress in the normal range and increase contractility allowing the preservation of stroke volume, this occurs at the expense of increased filling pressures. Diastolic dysfunction with increased filling pressure lead to left atrial (LA) dilatation and significantly contributes to the development of symptoms.

Despite successful surgery, AS patients have increased long-term mortality and morbidity compared to the general population, and the outcome is largely determined by the degree of preoperative structural LV and LA alterations. This has led to the theory that AVR prior to the development of symptoms could improve outcome, a view supported by prospective and retrospective studies.These studies were however small, with some important limitations. In addition, there has been a concern that operative risk and prosthetic valve related long-term morbidity and mortality does not justify surgery on every asymptomatic patient with severe AS. Numerous studies have suggested that markers of LV structure and function, particularly LA volume index,E/e' and brain natriuretic peptides (BNP) all reflecting LV filling pressures may identify patients with benefit of early AVR. Accordingly, the most recent European guideline for management of valvular disease has implemented BNP as a class IIa recommendation for AVR in asymptomatic AS patients,although no randomized studies have demonstrated that early surgery based on these markers improve prognosis.

The purpose of this study is thus to evaluate if early AVR in patients with signs of elevated LV filling pressuresmay improve long-term outcome in patients with asymptomatic severe AS, compared to conventional symptom-guided surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Severe AS defined as

  1. aortic valve area (AVA) ≤1 cm2, AND
  2. Transvalvular maximum velocity (Vmax) ≥3.5 m/s AND
  3. AS severity evaluated severe by a heart valve team conference. In cases where severity is not unambiguous an integrative approach will be utilized combining echocardiographic markers of valve severity and LV function, and if necessary aortic valve calcification estimated by non-contrast CT.

     2. Considered to be asymptomatic (estimated by a consultant in cardiology) 3. Considered to be candidate for AVR (transcatheter AVR/surgical AVR) 4. Sign of increased LV filling pressures18 or reduced longitudinal LV systolic function

  <!-- -->

  1. Left atrial volume index (LAVi) > 34 ml/m2; OR
  2. ratio of early diastolic peak mitral inflow velocity (E) to early mitral annulus diastolic velocity (e') ratio E/e'avg>13; OR
  3. Threefold elevation in NT-proBNP compared to the upper expected age and gender value. OR
  4. GLS>-15 5. Age ≥18 years 6. Signed informed consent

Exclusion Criteria:

1. LVEF<50%
2. Very severe AS defined as Vmax>5 m/s.
3. Concomitant severe valvular disease other than AS
4. Previous valvular surgery
5. Estimated glomerular filtration rate<30 ml/min/m2
6. Dementia
7. Women of childbearing potential
8. Inability to provide informed consent
9. Age>85 years.
10. Supravalvular or subvalvular AS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | After 379 events (approx 5 years)
  All-cause mortality assessed by Danish patient records

SECONDARY OUTCOMES:
Combined endpoint | After 379 events (approx 5 years)
  All-cause mortality + hospitalization due to heart failure and stroke
all-cause mortality in patients with low-gradient AS | After 379 events (approx 5 years)
  All-cause mortality in patients with meangradient <40 mmHg
Combined endpoint in low-gradient AS | After 379 events (approx 5 years)
  All-cause mortality + hospitalization to heart failure and stroke when MG<40 mmHg

OTHER OUTCOMES:
Pericardiocentesis | 5 years
  Need of pericariocentesis
sternal infection | 5 years
  hospitalization due to sternal infection
Persistent renal failure | 5 years
  complete loss of renal function exceeding 4 weeks.
endocarditis | 5-years
  hospitalization due to endocarditis
major bleeding | 5 years
  intracerebral bleeding or bleeding resulting in substantial hemodynamic compromise requiring treatment instability

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: No